CLINICAL TRIAL: NCT05699330
Title: Subgenual Cingulate Deep Brain Stimulation for Apathetic Behavioral Variant Frontotemporal Dementia - A Pilot Trial
Brief Title: Subgenual Cingulate Deep Brain STIMulation for Apathetic Behavioral Variant FRONtotemporal Dementia
Acronym: FRONSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, University Professor, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-6126
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Frontotemporal Dementia; Deep Brain Stimulation
Keywords: Subgenual cingulate; Deep brain stimulation; Apathy; Behavioral variant
MeSH Terms: conditions — Frontotemporal Dementia; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral subgenual cingulate deep brain stimulation (SGC DBS) (Experimental): Deep Brain Stimulation (DBS) is a neurosurgical procedure involving the implantation of deep brain electrodes, connected via a subcutaneous extension wire, to an implantable pulse generator (IPG, or 'battery') that is implanted below the collarbone. All patients will receive deep brain stimulation (DBS) targeting the subgenual cingulate (SGC) bilaterally. No other changes to pre-existing treatment will be made. This is the only arm in this experiment.
  Interventions: Device: Bilateral subgenual cingulate deep brain stimulation (SGC DBS)

INTERVENTIONS:
Device: Bilateral subgenual cingulate deep brain stimulation (SGC DBS) — Deep Brain Stimulation (DBS) is a neurosurgical procedure involving the implantation of deep brain electrodes, connected via a subcutaneous extension wire, to an implantable pulse generator (IPG, or 'battery') that is implanted below the collarbone. All patients will receive deep brain stimulation (DBS) targeting the subgenual cingulate (SGC) bilaterally. No other changes to pre-existing treatment will be made. This is the only arm in this experiment.

SUMMARY:
Frontotemporal dementia (FTD), the most common dementia in individuals younger than 60 years of age, has no disease-modifying treatment. Neuroimaging studies have revealed salience and default mode network dysfunction, frontotemporal atrophy and hypometabolism as pathophysiological hallmarks of behavioral variant FTD (bvFTD). A key brain structure affected by bvFTD is the subgenual cingulate (SGC), which serves as a hub for multi-axonal projections to and from the ventromedial prefrontal, dorsal anterior cingulate, orbitofrontal, and dorsolateral frontal cortices, and limbic structures.

The disruption of these SGC projections in bvFTD result in the core clinical features of apathy, disinhibition, loss of empathy, compulsivity, hyperorality and loss of executive function. The central goal of this proposal is to use deep brain stimulation (DBS) for modulation of the SGC downstream projections to treat bvFTD. Investigators hypothesize that SGC DBS will drive activity in the dysfunctional networks, reverse hypometabolism, and potentially improve symptoms. To determine the physiologic effects and mechanisms of SGC DBS, investigators will assess cerebral metabolism by FDG-PET, connectivity by rsfMRI and MEG, atrophy by volumetric MRI, and neurodegenerative and neuroinflammatory biomarkers. The safety and preliminary efficacy data obtained in these patients will inform the possible future role of DBS in apathetic bvFTD.

DETAILED DESCRIPTION:
Study Design:

This is a single-center prospective, open-label, non-blinded, non-randomized, pilot study designed to evaluate the safety of deep brain stimulation (DBS) of the subgenual cingulate (SGC) in subjects diagnosed with apathetic behavioral variant frontotemporal dementia (abvFTD). In addition, the physiological and clinical effects of DBS will be assessed by neuroimaging and neuropsychological testing.

Investigators hypothesize that:

1. Bilateral subgenual cingulate deep brain stimulator implantation will be well-tolerated in apathetic behavioral variant frontotemporal dementia patients. In AIM 1 investigators will assess the safety of SGC DBS, by monitoring intraoperative and postoperative adverse events related to surgery and stimulation in abvFTD patients.
2. Bilateral subgenual cingulate deep brain stimulation will modulate brain circuits that are dysfunctional in patients with apathetic behavioral variant frontotemporal dementia. In AIM 2 investigators will determine the physiological impact and mechanisms of action of SGC DBS in abvFTD, by assessing cerebral metabolism with ¹⁸F-fluorodeoxyglucose (¹⁸F-FDG) PET scans, functional connectivity with magnetoencephalography and resting state functional magnetic resonance imaging, cerebral atrophy with volumetric MRI, and plasma and cerebrospinal fluid biomarkers of neurodegeneration (glial fibrillar acidic protein and neurofilament light chain) and neuroinflammation (Olink inflammation panels I and II) in abvFTD patients.
3. Bilateral subgenual deep brain stimulation may improve some of the six core clinical features of behavioral variant frontotemporal dementia. In AIM 3 investigators will assess the clinical consequences of SGC DBS abvFTD, by performing the following neuropsychological tests: Neuropsychiatric index (NPI) and Apathy Evaluation Scale - Clinician version (AES-C) for apathy, NPI for disinhibition, compulsivity and hyperorality; Interpersonal reactivity index (IRI) for loss of empathy; National Institutes of Health - Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (NIHEXAMINER) and Trail making test - A and B (TMT) for executive function; Social Cognition and Emotional Assessment (SEA)/Mini-SEA), and Frontotemporal lobar degeneration-modified Clinical Dementia Rating-I (FTLD CDR-I) for cognitive impairment.

Experimental Approach:

Investigators propose a 3-year open-label, single-arm, phase I study of subgenual cingulate deep brain stimulation for apathetic behavioral variant frontotemporal dementia. In years 1-2 investigators will screen frontotemporal dementia patients and enrol a total of 6 subjects who meet the study inclusion criteria. Prior to SGC DBS surgery, the subjects will undergo baseline neuroimaging (FDG PET, rsfMRI, MEG, vMRI and tractography), measurement of plasma and neuroinflammation (multiplex proximity extension assay (PEA) technology using Olink Explore Inflammation I and II panels), optional lumbar puncture (according to patient preference) for CSF biomarkers of neurodegeneration (GFAP) and NfL assays), and neuropsychological testing (NPI, AES-C, IRI, NIH-EXAMINER, TMT, SEA/mini-SEA and FTLD CDR-I). At 2 weeks after surgery, the DBS device will be turned on, with subsequent programming sessions at 4 weeks, 6 weeks, 8 weeks, 10 weeks, 3 months, 6 months, 9 months, 12 months and 24 months post-DBS surgery to optimize therapy. During programming, the DBS stimulation parameters will be titrated with the patient's apathy score, measured by AES-C, which is a validated 18-item apathy scale that can be easily administered in 10-20 minutes during the programming session. Full neuropsychological testing (NPI, AES-C, IRI, NIH-EXAMINER, TMT, SEA/mini-SEA and FTLD CDR-I ) will be performed at baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery. Measurement of plasma neuroinflammatory biomarkers (Olink inflammation panels I and II) will be done at baseline before DBS surgery, and at 3-months, 6-months, 9-months, 12-months and 24-months post-DBS surgery. Lumbar puncture to obtain CSF for biomarkers of neurodegeneration (GFAP and NfL) will be optional and will be offered at baseline before DBS surgery and at 12-months and 24-months post-DBS surgery. Neuroimaging studies (FDG PET, rsfMRI, MEG, and vMRI) will be done at baseline before DBS surgery, and at 6-months, 12-months and 24-months post-DBS surgery. The baseline assessments and postoperative follow up will take place at Toronto Western Hospital. Investigators anticipate to complete patient follow-up by the end of year 3. However, it is possible that the 24-month follow up of a few patients may extend into year 4, depending on when their DBS surgery is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 40-85 years
2. Diagnosis of image-supported behavioral variant frontotemporal dementia according to NIC-FTD and NACC FTLD guidelines
3. Apathy as one of the symptoms
4. Stable dose of baseline FTD medications for at least 3 months
5. The patient has an available caregiver or other appropriate knowledgeable informant who can reliably report on daily activities and function. The patient must also have a substitute decision maker, if different from caregiver, to sign the informed consent for participation in the study.

Exclusion Criteria:

1. Meets diagnostic criteria for other psychiatric diagnosis
2. Has other major Central Nervous System (CNS) disease that impairs motor, sensory or cognitive
3. Alcohol or illegal substance dependence within last 12 months
4. Other medical conditions which render anesthesia and surgery as unsafe as determined by neurosurgeon
5. Contraindications for MRI scanning, including implanted metallic devices (e.g., non-MRI-safe cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces.
6. Has a medical condition requiring a repetitive MRI body scan
7. Requires chemotherapy for the treatment of malignancy or requiring chronic oral or intravenous (immunosuppressive or) steroid therapy
8. Is unable to comply with study visit schedule and timeline
9. Past significant intracranial surgery
10. A female lactating or of child-bearing potential, with a positive pregnancy test or not using adequate contraception.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 24 months
  Patients will be closely monitored for adverse events following DBS surgery with regular check-ups at 3-months, 6-months, 12-months and 24-months post-DBS surgery

SECONDARY OUTCOMES:
Apathy Evaluation Scale - Clinician version (AES-C) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  Patients will regularly complete the 18-item AES-C to assess apathy at baseline and at follow up. The scores range from 18-72, with a score greater than 34 indicating apathy
Neuropsychiatric index (NPI) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  At follow up, patients will regularly complete the NPI questionnaire, which assesses 12 domains of behavioral disturbances in dementia. The severity scale has scores ranging from 1 to 3 points (1=mild; 2=moderate; and 3=severe) and the scale for assessing caregiver distress has scores ranging from 0 to 5 points (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=extreme distress).
Interpersonal reactivity index (IRI) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  Patients will regularly complete the IRI questionnaire at follow up. The IRI consists of 28-items answered on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales, each made up of 7 different items.
National Institutes of Health - Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (NIH-EXAMINER) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  At follow up, patients will regularly complete the NIH-EXAMINER battery, which generates 4 composite scores to measure overall executive dysfunction, cognitive control, working memory, and fluency.
Trail making test - A and B (TMT) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  At follow up, patients will regularly undergo the rail making tests, which measure the cognitive domains of processing speed, sequencing, mental flexibility and visual-motor skills and executive function. A cut-off time of 300 seconds is generally used to discontinue test administration and is therefore the typical maximum score.
Social Cognition and Emotional Assessment (SEA)/Mini-SEA) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  At follow up, patients will regularly undergo the SEA/Mini-SEA battery. The Social Cognition and Emotional Assessment (SEA) is designed to provide an overview of social cognition and other processes mediated by the orbital and medial frontal regions in people with frontotemporal dementia. It comprises five subtests (Max total score = 55).
Frontotemporal lobar degeneration-modified Clinical Dementia Rating-I (FTLD CDR-I) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  At follow up, patients will regularly complete the FTLD CDR-I questionnaire, which is the classic six-domain CDR plus two domains (behavior and language), specific for FTLD. A rating of "0" indicates normal behavioral or language status, while ratings of "1," "2," and "3" denote mild, modest, and severe deficits, respectively.
Plasma neuroinflammatory biomarkers (Olink inflammation panels I and II) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  Plasma will be obtain at follow up and used to measure neuroinflammatory biomarkers using the Olink inflammation panels I and II.
Cerebrospinal fluid biomarkers of neurodegeneration (GFAP and NfL) | Baseline before DBS surgery and at 12-months and 24-months post-DBS surgery
  Collection of cerebrospinal fluid by lumbar puncture will be optional. If a patient consents to have a lumbar puncture, cerebrospinal fluid will be obtained to measure biomarkers of neurodegeneration (GFAP and NfL).
Neuroimaging studies (FDG PET, rsfMRI, MEG, and vMRI) | Baseline before DBS surgery, and at 6-months, 12-months and 24-months post-DBS surgery
  Advanced neuroimaging (FDG PET, rsfMRI, MEG, and vMRI) will be done at baseline and follow up to check for cerebral glucose metabolism, connectivity and cerebral atrophy.
Free and Cued Selective Reminding Test (FCSRT) | Baseline before DBS surgery, and at 3-months, 6-months, 12-months and 24-months post-DBS surgery
  At follow up, patients will regularly complete the FCSRT, which is a multi-trial memory test that uses a "selective reminding" paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Lozano, MD, PhD, Principal Investigator — University Health Network, Toronto; Carmela Tartaglia, MD, Principal Investigator — University Health Network, Toronto; Cletus Cheyuo, MD, PhD, Study Director — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada